CLINICAL TRIAL: NCT05233358
Title: HAIC Combined With Second-line "Target Immunity" for Advanced Hepatocellular Carcinoma With Low Response or Failure of TACE Combined With First-line "Target Immunity": A Prospective, Randomized- Control, Multicenter Clinical Trial
Brief Title: HAIC Combined With Second-line "Target Immunity" for HCC With TACE Standard Treatment Low Response or Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Central Hospital of Lishui City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZJLS-KLDMIR-22001
Record Dates: First submitted 2022-01-24; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Hepatic Artery Infusion Chemotherapy; Transarterial Chemoembolization; Target Immunity; Advanced
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — regorafenib; Immune Checkpoint Inhibitors; camrelizumab; sintilimab; Nivolumab; pembrolizumab; toripalimab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAIC combined with regorafenib and immune checkpoint inhibitors (Experimental): Subjects received FOLFOX regimen HAIC treatment, within 2 weeks of regorafenib (28 days as a cycle, 80-160 mg qd regorafenib orally on days 1-21) and immune checkpoint inhibitors (continue treatment according to the original plan, 1 cycle every 3 weeks) treatment. HAIC treatment was repeated every 3 weeks for a maximum of six cycles.
  Interventions: Procedure: Hepatic Artery Infusion Chemotherapy; Drug: Regorafenib; Drug: Immune Checkpoint Inhibitors
- TACE combined with regorafenib and immune checkpoint inhibitors (Active Comparator): Choose traditional precise cTACE or dTACE treatment, and receive regorafenib within 2 weeks (28 days as a cycle, 80-160mg qd regorafenib orally on d1-21) and immune checkpoint inhibitors (continue treatment according to the original plan, every 3 weeks as a cycle) treatment. CT or MRI examination was repeated 4-6 weeks after the operation to evaluate whether there were active lesions. If there were still active lesions, one repeat TACE could be performed, and the number of TACE was less than 3 times.
  Interventions: Procedure: Transarterial Chemoembolization; Drug: Regorafenib; Drug: Immune Checkpoint Inhibitors

INTERVENTIONS:
Procedure: Hepatic Artery Infusion Chemotherapy — HAIC adopts FOLFOX chemotherapy regimen, hepatic arteriography through a radial artery or femoral artery cannulation, routine hepatic artery cannulation, imaging, infusion of chemotherapy drugs into hepatic artery: oxaliplatin 85 mg/m2 on the first day for 0-3 hours, folinic acid 400 mg/m2 for 3-4.5 hours on day 1, fluorouracil 400 mg/m2 for 4.5-6.5 hours on day 1, and fluorouracil 2500 mg/m2 for 46 hours on days 1-3.
  Other Names: HAIC
  Arms: HAIC combined with regorafenib and immune checkpoint inhibitors
Procedure: Transarterial Chemoembolization — Treatment regimens have chosen "lipiodol-based" hepatic arterial chemoembolization, with lipiodol dosage varying from 5-20ml depending on tumor size. The chemotherapy drug is gemcitabine 1.0 combined with 100mg oxaliplatin, combined with 1/3 to 1 dose of solid embolic agent (the dosage is determined by the investigator based on the tumor size). After uniform emulsification, the drug is injected into the supplying blood vessels and stops when the intravascular blood flow is slow. Later, angiography is performed again, and the tumor staining disappears and the supplying artery is occlusions.
  CT or MRI scans are performed 4 to 6 weeks postoperatively to assess the presence of active lesions. Repeat TACE if active lesions are still present. The frequency of TACE treatment is determined by the investigator and is given according to the patient's condition, generally 2-4 times. The interval between TACE treatments is 30-45 days, with a maximum of six cycles.
  Other Names: TACE
  Arms: TACE combined with regorafenib and immune checkpoint inhibitors
Drug: Regorafenib — Regorafenib is administered for 28 days per treatment cycle, with oral regorafenib on days 1-21, 80-160 mg once daily. The dose is adjusted according to adverse reactions, with a minimum of 80 mg.
  Other Names: second-line target drug
Drug: Immune Checkpoint Inhibitors — Optional immune checkpoint inhibitors include Camrelizumab, Sintilimab, Nivolumab, Pembrolizumab, and Toripalimab. Treatment is based on the immune checkpoint inhibitor before the patients are randomized into the group, and it is not recommended to replace the immune checkpoint inhibitor. The dosage is 200 mg, intravenous infusion, D1, once every 21 days (Q3W). Dosing interruption or dose reduction may be necessary based on individual safety and tolerability considerations; dosing with immune checkpoint inhibitors should not be suspended for more than 4 weeks.
  Other Names: Camrelizumab, Sintilimab, Nivolumab, Pembrolizumab, Toripalimab

SUMMARY:
This study is a prospective, randomized controlled, multicenter clinical study. The purpose of this study is to explore the efficacy and safety of hepatic artery infusion chemotherapy (HAIC) combined with second-line regorafenib and immune checkpoint inhibitors in the treatment of transarterial chemoembolization (TACE) combined with first-line molecular targeted drugs and immune checkpoint inhibitors with low response or failure in advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
This is a randomized, open, parallel-controlled, multi-center clinical trial with a type of comparison using a merit test. This study will recruit 176 patients with advanced liver cancer who have received TACE combined with first-line "target immune" therapy and were rated as low response or treatment failure according to mRECIST criteria in multiple research centers across the country. Subjects randomly assigned to the experimental group will receive HAIC in combination with regorafenib and immune checkpoint inhibitors, and subjects randomly assigned to the control group will receive TACE in combination with regorafenib and immune checkpoint inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in this study and sign the informed consent;
* Age ≥18 years old to 70 years old;
* Patients diagnosed with primary liver cancer by histopathology, cytology or imaging;
* The China liver cancer staging is IIb-IIIa;
* Patients with intermediate and advanced liver cancer who must receive at least one cycle of TACE combined with first-line "target immune" therapy and are assessed as partial remission (PR), stable disease (SD）(low response), and progressive disease (PD) (failure) according to mRECIST criteria;
* At least one measurable (based on RECIST 1.1 criteria and mRECIST criteria) lesions, tumor lesions located at the local treatment site, if progressed, considered measurable;
* Local treatment (surgery, radiotherapy, radiofrequency/microwave ablation, cryoablation, percutaneous ethanol injection) can be used in the past, but it must be completed before 3 months;
* ECOG PS score ≤ 2;
* Child-Pugh liver function classification: grade A/B (≤9 points);
* Expected survival > 3 months;
* Patients with active hepatitis B virus (HBV) infection: HBV DNA ≤2000 IU/mL (104 cps/ml) obtained within 28 days prior to initiation of study treatment, and receiving anti-HBV treatment for at least 14 days prior to study entry (based on local standard treatment) and willing to continue to receive treatment during the study;

Exclusion Criteria:

* Have received HAIC treatment in the past;
* Known allergy to possible therapeutic drugs;
* Previously received regorafenib treatment;
* According to the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0), the toxicity grade caused by TACE combined with first-line "target immunity" treatment is > grade 3;
* Patients with liver decompensation, including esophageal or gastric variceal bleeding or hepatic encephalopathy, pregnancy or breastfeeding and other aggressive malignant diseases;
* Use immunosuppressive drugs and high-dose hormone therapy within 2 weeks before randomization to achieve the purpose of immunosuppression (dose>10mg/day prednisone or other hormones with equivalent efficacy);
* CART treatment within 3 months before randomization;
* Laboratory test values 1 week before randomization: blood routine: ① leukocyte <3.0×109/L; ② absolute neutrophil count <1.5×109/L; ③ platelets <75×109/L; ④ hemoglobin < 90g/L; liver function: ①serum albumin<30g/L; ②ALT and AST>5×ULN; renal function: ①serum creatinine>1.5×ULN; ②Cr clearance rate<50ml/min; ③estimated renal small Globular filtration rate (eGFR) <30 mL/min/1.73 m2; coagulation function: ① international normalized ratio (INR)> 2; ② prothrombin time (PT) exceeding the range of normal control> 6 seconds;
* Uncontrolled hypertension (systolic blood pressure > 180 mmHg, diastolic blood pressure > 110 mmHg);
* Uncontrollable diabetes;
* Active heart disease, including myocardial infarction, unstable angina pectoris, NYHA class II and above heart failure, and poorly controlled arrhythmias (including QTcF interval >450 ms in men and >470 ms in women);
* Women are pregnant or breastfeeding;
* History of any active autoimmune disease or autoimmune disease, including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, vasculitis, glomerulonephritis, hyperthyroidism, or hypothyroidism, asthma requiring bronchodilator treatment, etc;
* Uncontrolled clinically significant ascites (uncontrolled with diuretics or paracentesis);
* Combined with active infection, except HBV and HCV;
* Arterial or venous thrombosis or embolic events, such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis or pulmonary embolism, occurred 6 months before starting drug treatment;
* Known central nervous system (CNS) metastasis or meningeal metastasis;
* The patient cannot receive follow-up or is participating in other clinical trials;
* The investigator believes that the patient has other conditions that make it inappropriate to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | The time from enrollment to tumor progression or death from any cause, whichever came first, measured in "months", assessed up to 2 years.
  The 6-month, 1-year and 2-year progression-free survival rates were evaluated.

SECONDARY OUTCOMES:
Overall Survival | Time from enrollment to death from any cause, in "months", assessed up to 2 years. For patients who are still alive at the time of data analysis, overall survival is calculated based on the date when the patient is last known to be alive.
  The survival rates were evaluated.
To Tumor Untreatable Progression | The time interval between receiving HAIC or TACE and the patient's inability to receive further intra-arterial treatment, assessed up to 12 months.
  End point of antitumor drug trial.
Objective Response Rate | Proportion of patients who achieved complete remission (CR) or partial remission (PR) according to mRECIST criteria, assessed up to 12 months.
  The 1-, 3-, 6-, and 12 months ORR were evaluated.
Disease Control Rate | Proportion of patients with complete remission (CR), partial remission (PR), and stable disease (SD) according to mRECIST criteria, assessed up to 12 months.
  The 1-, 3-, 6-, and 12 months DCR were evaluated.
Duration of Overall Response | The time from the first assessment of the tumor as complete remission or partial remission to the first assessment as disease progression or death from any cause, assessed up to 12 months.
  Evaluation index of clinical efficacy of anticancer drugs.
The incidence of adverse events and serious adverse events | Every follow-up time, assessed up to 2 years.
  Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Liyun Zheng, MD., Study Director — The Central Hospital of Lishui City

IPD SHARING:
Plan to Share IPD: Yes
Statistical analysis plan, informed consent form, and clinical study report can be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within six months after the trial is completed.
Access Criteria: Shared data is not available for downloading, but can only be browsed. To download the data, you must contact the researchers. Shared data does not provide any private information of the participants.

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Finn RS, Ikeda M, Zhu AX, Sung MW, Baron AD, Kudo M, Okusaka T, Kobayashi M, Kumada H, Kaneko S, Pracht M, Mamontov K, Meyer T, Kubota T, Dutcus CE, Saito K, Siegel AB, Dubrovsky L, Mody K, Llovet JM. Phase Ib Study of Lenvatinib Plus Pembrolizumab in Patients With Unresectable Hepatocellular Carcinoma. J Clin Oncol. 2020 Sep 10;38(26):2960-2970. doi: 10.1200/JCO.20.00808. Epub 2020 Jul 27. PMID 32716739
- [Background] Zhu AX, Finn RS, Edeline J, Cattan S, Ogasawara S, Palmer D, Verslype C, Zagonel V, Fartoux L, Vogel A, Sarker D, Verset G, Chan SL, Knox J, Daniele B, Webber AL, Ebbinghaus SW, Ma J, Siegel AB, Cheng AL, Kudo M; KEYNOTE-224 investigators. Pembrolizumab in patients with advanced hepatocellular carcinoma previously treated with sorafenib (KEYNOTE-224): a non-randomised, open-label phase 2 trial. Lancet Oncol. 2018 Jul;19(7):940-952. doi: 10.1016/S1470-2045(18)30351-6. Epub 2018 Jun 3. PMID 29875066
- [Background] Odagiri N, Hai H, Thuy LTT, Dong MP, Suoh M, Kotani K, Hagihara A, Uchida-Kobayashi S, Tamori A, Enomoto M, Kawada N. Early Change in the Plasma Levels of Circulating Soluble Immune Checkpoint Proteins in Patients with Unresectable Hepatocellular Carcinoma Treated by Lenvatinib or Transcatheter Arterial Chemoembolization. Cancers (Basel). 2020 Jul 24;12(8):2045. doi: 10.3390/cancers12082045. PMID 32722224
- [Background] Wang Y, Zhou C, Liu J, Shi Q, Huang S, Yang C, Li T, Chen Y, Xiong B. Increased Liquefactive Necrosis Formation After Transarterial Chemoembolization Combined with Molecular Targeted Agents Plus Immune Checkpoint Inhibitors for Hepatocellular Carcinoma. Cancer Manag Res. 2021 Sep 7;13:6935-6941. doi: 10.2147/CMAR.S328812. eCollection 2021. PMID 34522136
- [Background] Li J, Qin S, Xu R, Yau TC, Ma B, Pan H, Xu J, Bai Y, Chi Y, Wang L, Yeh KH, Bi F, Cheng Y, Le AT, Lin JK, Liu T, Ma D, Kappeler C, Kalmus J, Kim TW; CONCUR Investigators. Regorafenib plus best supportive care versus placebo plus best supportive care in Asian patients with previously treated metastatic colorectal cancer (CONCUR): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2015 Jun;16(6):619-29. doi: 10.1016/S1470-2045(15)70156-7. Epub 2015 May 13. PMID 25981818
- [Background] Bruix J, Qin S, Merle P, Granito A, Huang YH, Bodoky G, Pracht M, Yokosuka O, Rosmorduc O, Breder V, Gerolami R, Masi G, Ross PJ, Song T, Bronowicki JP, Ollivier-Hourmand I, Kudo M, Cheng AL, Llovet JM, Finn RS, LeBerre MA, Baumhauer A, Meinhardt G, Han G; RESORCE Investigators. Regorafenib for patients with hepatocellular carcinoma who progressed on sorafenib treatment (RESORCE): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Jan 7;389(10064):56-66. doi: 10.1016/S0140-6736(16)32453-9. Epub 2016 Dec 6. PMID 27932229
- [Background] Ikeda M, Shimizu S, Sato T, Morimoto M, Kojima Y, Inaba Y, Hagihara A, Kudo M, Nakamori S, Kaneko S, Sugimoto R, Tahara T, Ohmura T, Yasui K, Sato K, Ishii H, Furuse J, Okusaka T. Sorafenib plus hepatic arterial infusion chemotherapy with cisplatin versus sorafenib for advanced hepatocellular carcinoma: randomized phase II trial. Ann Oncol. 2016 Nov;27(11):2090-2096. doi: 10.1093/annonc/mdw323. Epub 2016 Aug 29. PMID 27573564